CLINICAL TRIAL: NCT00582673
Title: A Multi-centre, Randomized, Double-blind, Placebo Controlled, Parallel-group, Multiple Oral Dose Titration Study in Patients With Parkinson's Disease to Assess the Efficacy of AFQ056 in Reducing L-dopa Induced Dyskinesias, and the Safety and Tolerability of AFQ056 in Combination With L-dopa
Brief Title: Efficacy and Safety of AFQ056 in Reducing L-dopa Induced Dyskinesias in Parkinson's Disease Patients, and Safety in Combination With L-dopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAFQ056A2203
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's, L-dopa, dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AFQ056
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of administration of AFQ056 in combination with L-dopa, in reducing the number of L-dopa related dyskinesias in Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease
* Patients with L-dopa induced dyskinesia for at least 3 months
* Patients with L-dopa treatment for at least 3 years, stable for 1 month minimum

Exclusion Criteria:

* History of severe allergy to food or drugs
* Very low or high body weight.
* Prior surgery for Parkinson's Disease
* Smokers

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number and severity of Dyskinesias and the safety and tolerability of administering AFQ056 in combination with L-dopa | throughout the study

SECONDARY OUTCOMES:
Number and severity of Dyskinesias and the safety and tolerability of administering AFQ056 in combination with L-dopa | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigative site
Locations (5):
- Germany (5):
  - Novartis Investigator Site, Dresden
  - Novartis Investigator Site, Kassel
  - Novartis Investigator Site, Leun
  - Novartis Investigator Site, Marburg
  - Novartis Investigator Site, Tübingen

REFERENCES:
- [Derived] Berg D, Godau J, Trenkwalder C, Eggert K, Csoti I, Storch A, Huber H, Morelli-Canelo M, Stamelou M, Ries V, Wolz M, Schneider C, Di Paolo T, Gasparini F, Hariry S, Vandemeulebroecke M, Abi-Saab W, Cooke K, Johns D, Gomez-Mancilla B. AFQ056 treatment of levodopa-induced dyskinesias: results of 2 randomized controlled trials. Mov Disord. 2011 Jun;26(7):1243-50. doi: 10.1002/mds.23616. Epub 2011 Apr 11. PMID 21484867